CLINICAL TRIAL: NCT00617474
Title: The Effect of Erythropoietin Usage in Renal Function After Kidney Transplantation, in Early Phase, in Contrast to Placebo Group
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Labbafinejhad Hospital (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr.Poorrezagholi, Shaheed Beheshti Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L1386; 200786
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Transplantation, Kidney
Keywords: erythropoietin; kidney allograft survival; Recombinant Erythropoietin; erythropoietin (Epo)-induced protein 29, human
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Group of patient with anemia, that treated by erythropoietin
  Interventions: Drug: Erythropoietin
- 2 (Placebo Comparator): Patients group with anemia that treated by placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythropoietin — sub cutaneous injection, 2000 unit in per injection, 3 times 1 week.
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
The study hypothesis is that erythropoietin usage after kidney transplantation, in early phase, can improve the outcome for patients and their graft increasing patient and graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Hb: >8 and <10 gr/dl
* Age: >18 and <55 years
* Cholesterol: <300 mg/dl
* Triglyceride: <400 mg/dl
* First Transplantation
* Protocol of Immunosuppression: CSA + MMF + Prednisolone
* Systolic BP: <14
* Diastolic BP: <9

Exclusion Criteria:

* History of specified cardiac disease
* Second Transplantation or more
* Hb: <7gr/dl
* The patient needs to infusion of blood
* Evidence of local or systemic infection, at the time of EPO injection
* Presence of ATN / DGF after transplantation
* Presence of emergent hypertension
* High risk patients ( Like; PRA>50%)
* Past history of hypersensitivity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-09 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
We will study the well-being of renal function by evaluation of plasma Cr,GFR,PTDA scan & biopsy proven(If it is necessary to prove the rejection)about measuring of patient - graft survival. | May,2008